CLINICAL TRIAL: NCT04095637
Title: A Prospective Randomised Control Trial of Mako Medial Unicondylar Knee Arthroplasty Versus Jig-based Oxford Unicompartmental Knee Arthroplasty With Navigation Contro
Brief Title: RCT: Mako Medial Unicondylar Knee Arthroplasty vs Oxford Unicondylar Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Stryker Instruments (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16/0773
Record Dates: First submitted 2019-07-17; First posted 2019-09-19 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Unicompartmental Knee Replacement; Osteo Arthritis Knee; Surgery
Keywords: alignment; computer navigation; implant position; mako robot; makoplasty; unicondylar knee replacement

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Mako medial UKA (Experimental): Mako medial unicondylar knee arthroplasty
  Interventions: Device: Medial knee arthroplasty
- Oxford media UKA (Active Comparator): Oxford unicompartmental knee arthroplasty with navigation control
  Interventions: Device: Medial knee arthroplasty

INTERVENTIONS:
Device: Medial knee arthroplasty — Surgical intervention where the medial portion of the knee is replaced by an artificial metal and polyethylene implant

SUMMARY:
The overall aim of this prospective, randomised, single-blinded, controlled trial is to compare clinical outcomes and accuracy of implant positioning in Mako robotic UKA versus jig-based Oxford UKA with navigation control. Patients receiving the Mako robotic UKA (Stryker Ltd) will form the investigation group and those undergoing the jig-based Oxford UKA (Zimmer-Biomet Ltd) with navigation control will form the control group.

The primary objective in this study is to compare accuracy of component positioning as assessed by postoperative low radiation dose CT scan between conventional Jig-based Oxford UKA with navigation control and Mako robotic UKA.

ELIGIBILITY:
Inclusion Criteria:

* • Patient has medial unicompartmental knee osteoarthritis requiring primary UKA

  * Patient and Surgeon are in agreement that UKA is the most appropriate treatment
  * Patient is fit for surgical intervention following review by surgeon and anaesthetist
  * Patient is between 40-80 years of age at time of surgery
  * Gender: male and female
  * Patient must be capable of giving informed consent and agree to comply with the postoperative review program
  * Patient must be a permanent resident in an area accessible to the study site
  * Patient must have sufficient postoperative mobility to attend follow-up clinics and allow for radiographs to be taken

Exclusion Criteria:

* • Patient is not suitable for primary UKA e.g. multi-compartmental knee osteoarthritis, anterior cruciate ligament rupture

  * Patient is not medically fit for surgical intervention
  * Patient requires revision surgery following previously failed correctional osteotomy or ipsilateral UKA
  * Patient is immobile or has another neurological condition affecting musculoskeletal function
  * Patient is less than 40 years of age or greater than 80 years of age
  * Patient is already enrolled on another concurrent clinical trial
  * Patient is unable or unwilling to sign the informed consent form specific to this study
  * Patient is unable to attend the follow-up programme
  * Patient is non-resident in local area or expected to leave the catchment area postoperatively

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-11-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of component positioning | 6 weeks post-op
  Comparison of accuracy of component positioning as assessed by postoperative low radiation dose CT scan

SECONDARY OUTCOMES:
Lower limb alignment | Pre-op then 6 weeks, 6 months, 1 and 2 years post-op
  Lower limb alignment in the coronal, axial, and sagittal planes as assessed by postoperative low radiation dose CT scan at 6 weeks after surgery.
Femoral implant alignment | Pre-op then 6 weeks, 6 months, 1 and 2 years post-op
  Femoral implant alignment in the coronal, axial, and sagittal planes as assessed by postoperative low radiation dose CT scan at 6 weeks after surgery.
Tibial implant alignment | Pre-op then 6 weeks, 6 months, 1 and 2 years post-op
  Tibial implant alignment in the coronal, axial, and sagittal planes as assessed by postoperative low radiation dose CT scan at 6 weeks after surgery.
Operating time | Intraoperative
  Length of time of operation in minutes
Time to discharge | 6 weeks post op
  Length of hospital admission from admission date to documented discharge from hospital
Oxford Knee Score (OKS) | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure via questionnaire; cumulative score with best being 48, worst being 0
Short form SF-12 | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure via questionnaire; cumulative score via 12 questions pertaining to perception of current physical and mental health; higher score best score, lower score worse score
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure via questionnaire; cumulative score with 0 being best score
Knee injury and Osteoarthritis Outcome Score (KOOS) Osteoarthritis Outcome Score (KOOS) | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Patient recorded outcome measure via questionnaire; 6 domains contribute to overall percentage; 100% being best score
European Quality of Life questionnaire with 5 dimensions for adults (EQ-5D) | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Health-related quality of life via 5 domains; score -1 to 1 with 1 being best score
Mobilisation distance (metres) | Pre-op; 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  How far patient can walk in metres
Use of mobility aids | Pre-op then 6 weeks post-op; 6 months post-op; 1 year post-op; 2 years post-op
  Documenting the use of any mobility aid to assist with ambulation; can include wheelchair, walker, crutches, sticks or no aid required
Range of movement | Pre-op then 6 weeks post-op, 6 months post-op, one year post-op; 2 years post-op
  Range of movement of knee joint in degrees, typically from 0 to 140 degrees; higher number is better score
Complications | during inpatient admission and postoperatively at 6- weeks, 6 months, 1 year and 2 years
  Complications as relating to surgery; to include pain; fracture; neurovascular injury; blood clots; infection of wound; infection of artificial joint; pain; heart attack; stroke; pulmonary embolus; return to operating theatre; revision surgery; death

CONTACTS AND LOCATIONS:
Overall Officials: Fares S Haddad, Study Chair — UCL Hospitals NHS Foundation Trust; Babar Kayani, Principal Investigator — UCL Hospitals NHS Foundation Trust
Locations (1):
- UCL Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Derived] Kayani B, Konan S, Tahmassebi J, Ayuob A, Moriarty PD, Haddad FS. Robotic-arm assisted medial unicondylar knee arthroplasty versus jig-based unicompartmental knee arthroplasty with navigation control: study protocol for a prospective randomised controlled trial. Trials. 2020 Aug 17;21(1):721. doi: 10.1186/s13063-020-04631-5. PMID 32807219